CLINICAL TRIAL: NCT03371745
Title: A Prospective, Randomized, Controlled Clinical Trial Evaluating the Superiority of Preimplantation Genetic Screening (PGS) and Deferred Transfer of Cryopreserved Embryos Over "Freeze-Only" Deferred Transfer Without PGS or Immediate Embryo Transfer During a "Fresh" In Vitro Fertilization Cycle
Brief Title: The PrISICE Clinical Trial (Pre-Implantation Screening and Investigation on the Cryopreservation of Embryos)
Acronym: PrISICE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The Reproductive Medicine Network was disbanded
Sponsor: Yale University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of California, San Francisco (Other); University of Pennsylvania (Other); Augusta University (Other); Penn State University (Other); University of North Carolina (Other); University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PrISICE
Record Dates: First submitted 2017-12-08; First posted 2017-12-13 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Cryopreservation; Embryo Transfer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PGS-FET (Active Comparator): The PGS-FET arm involves deferred transfer of embryos following cryopreservation at the blastocyst stage following pre-implantation genetic screening. This arm will culture embryos to day 5/6/7 (blastocyst stage). The embryos will be cryopreserved following trophectoderm biopsy. A subsequent frozen embryo transfer cycle will be performed during which 1 euploid (chromosomally normal) embryo will be thawed and transferred.
  Interventions: Procedure: Trophectoderm biopsy; Procedure: Cryopreservation; Procedure: Embryo Transfer
- FET (Active Comparator): The "Freeze only" arm involves the deferred transfer of embryos following cryopreservation. In this arm embryos will be cryopreserved. A subsequent frozen embryo transfer cycle will be performed during which one or more embryos will be thawed and transfered based on local clinical site, age-specific embryo number transfer guidelines.
  Interventions: Procedure: Cryopreservation; Procedure: Embryo Transfer
- Fresh (Active Comparator): The Fresh arm will have an immediate embryo(s) transfer based on local clinical site, age-specific embryo number transfer guidelines within the stimulation cycle.
  Interventions: Procedure: Embryo Transfer

INTERVENTIONS:
Procedure: Trophectoderm biopsy — Biopsy at blastocyst stage of trophectoderm cells for comprehensive evaluation of the eupolid status of the embryo.
  Arms: PGS-FET
Procedure: Cryopreservation — Rapid freezing using vitrification
  Arms: FET; PGS-FET
Procedure: Embryo Transfer — Transfer of embryo that has been cultured in vitro into the uterus

SUMMARY:
The trial objective is to determine whether the deferred transfer of embryos following cryopreservation at the blastocyst stage following pre-implantation genetic screening (PGS-FET) improves live birthrates compared to both the deferred transfer of cryopreserved embryos without PGS (FET) and immediate transfer at the conclusion of a "fresh" in vitro fertilization (IVF) cycle (Fresh). Additionally, whether "freeze-only" (FET) improves live birth rates compared to "fresh" will be determined.

DETAILED DESCRIPTION:
This will be a multi-center, prospective randomized clinical trial comparing three standards of care:

Group 1: PGS-FET group: deferred transfer of day 5/6/7 (blastocyst stage) embryos cryopreserved following trophectoderm biopsy Group 2: "freeze-only" (FET) group: deferred transfer of frozen/thawed embryos without biopsy Group 3: "fresh" ET group: immediate transfer of "fresh" embryos in the stimulation cycle.

1539 eligible couples will be recruited to participate. Couples will be randomized at retrieval to undergo cryopreservation with deferred embryo transfer, with or without PGS, or fresh embryo transfer during the cycle of egg retrieval. Number of embryos to transfer will be based on clinical estimation of embryo quality and will not exceed ASRM guidelines for embryo transfer number including newly revised guidelines. We are aware that the number of embryos transferred, to maintain enrollment, may not be equivalent, with likely more embryos transferred in patients not having PGS. The primary outcome of live birth/retrieval, with a secondary outcome of healthy singleton birth, may reflect the true benefit of PGS.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo in vitro fertilization for treatment of infertility (1st or 2nd "fresh" attempt); subject can have had no more than one prior failed "fresh" IVF cycle
* Couple able to participate in a research project

  * Able to understand study requirements
  * Willing to sign informed consent
  * Able to return for required follow-up
  * Access to telephone
  * Ability to read and write
* Normal uterine cavity evaluation within one year of enrollment

Exclusion Criteria:

* Medical conditions which may complicate treatment
* No plans to undergo embryo transfer
* Medical contraindication to the transfer of more than a single embryo (i.e. congenital uterine anomaly).
* Concurrent participation in any other interventional trial
* Recurrent pregnancy loss
* Known chromosomal abnormality (e.g. translocation)
* Pre-implantation genetic diagnosis requiring blastocyst biopsy

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-08-21 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Live Birth | up to 9 months or time of birth
  The number of subjects who deliver a live born infant which will be calculated into a live born delivery rate.

CONTACTS AND LOCATIONS:
Overall Officials: Esther Eisenberg, MD, Study Director — Eunice Kennedy Shriver National Institue of Child Health and Human Development; Nanette Santoro, MD, Study Chair — University of Colorado, Denver; Marcelle I Cedars, MD, Principal Investigator — University of California, San Francisco; Christos Coutifaris, MD PhD, Principal Investigator — University of Pennsylvania; Heping Zhang, PhD, Study Director — Yale University
Locations (3):
- United States (3):
  - University of California San Francisco, San Francisco, California
  - University of Oklahoma, Oklahoma City, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
IPD data will be deposited in DASH following publication of the results of the primary paper and when the deidentified data have been put into a format that is acceptable for DASH submission.
Time Frame: After publication of the results of the primary paper and when the de-identified data have been put into a format that is acceptable for DASH submission.

REFERENCES:
- [Derived] Cornelisse S, Zagers M, Kostova E, Fleischer K, van Wely M, Mastenbroek S. Preimplantation genetic testing for aneuploidies (abnormal number of chromosomes) in in vitro fertilisation. Cochrane Database Syst Rev. 2020 Sep 8;9(9):CD005291. doi: 10.1002/14651858.CD005291.pub3. PMID 32898291
- See also: Related Info — http://c2s2.yale.edu/rmn/